CLINICAL TRIAL: NCT02299739
Title: Liver Enzyme Abnormalities and Its Risk Factors in Taking Traditional Herbal Medicine in Korea
Brief Title: Liver Enzyme Abnormalities and Risk Factors in Taking Herbal Medicine
Status: Completed | Type: Observational
Sponsor: Jaseng Hospital of Korean Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: JS-CT-2013-02
Record Dates: First submitted 2014-11-18; First posted 2014-11-24 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Drug-Induced Liver Injury; Musculoskeletal Diseases
Keywords: Herbal Medicine; Complementary Therapies; Liver Function Tests; Risk Factors
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury; Musculoskeletal Diseases | interventions — Phytotherapy; Acupuncture Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Herbal medicine — Herbal medicine was taken 3 times daily in dried powder (2g) and water-base decoction form (120ml) (Ostericum koreanum, Eucommia ulmoides, Acanthopanax sessiliflorus, Achyranthes bidentata, Psoralea corylifolia, Peucedanum japonicum, Cibotium barometz, Lycium chinense, Boschniakia rossica, Cuscuta chinensis, and Atractylodes japonica).
  Other Names: Traditional herbal medicine
Procedure: Acupuncture — Acupuncture treatment was administered 1-2 times daily using mainly Ah-shi points and local acupuncture points.
Procedure: Pharmacopuncture — Select ingredients similar to those included in the oral herbal medicine (Ostericum koreanum, Eucommia ulmoides, Acanthopanax Sessiliflorus, Achyranthes bidentata, Psoralea corylifolia, Peucedanum japonicum, Cibotium barometz, Lycium chinense, Boschniakia rossica, Cuscuta chinensis, and Atractylodes japonica) were freeze dried into powder form after decoction, then diluted in normal saline and adjusted for acidity and pH to be used in injections. The pharmacopuncture injections were injected once daily to the amount of 1 cc and Ah-shi points and local acupuncture points (CPL, 1 cc, 26G x 1.5 syringe, Shinchang medical co., Korea).
Procedure: Bee venom pharmacopuncture — Bee venom pharmacopuncture was applied after confirming a negative reaction to the hypersensitivity skin test. Diluted bee venom (saline:bee venom ratio, 10,000:1) was injected at 4-5 acupoints at the physician's discretion. Each acupuncture point was injected with approximately 0.2 cc to a total of 0.5-1 cc using disposable injection needles (CPL, 1 cc, 26G x 1.5 syringe, Shinchang medical co., Korea).
Procedure: Chuna manipulation — Chuna was administered 3-5 times a week. Chuna is a Korean version of spinal manipulation that incorporates conventional spinal manipulation techniques for mobilization involving high-velocity, low amplitude thrusts to joints slightly beyond the passive range of motion and gentle force to joints within the passive range of movement.

SUMMARY:
Herb-induced liver injury is an important issue in musculoskeletal diseases where herbal medicine is most frequently used. The low prevalence of drug-induced liver injury (DILI) gives rise to the need for large-scale patient studies. We assessed the prevalence of liver injury of 6,894 musculoskeletal disease inpatients taking herbal medicine.

DETAILED DESCRIPTION:
Herb-induced liver injury is an important issue in musculoskeletal diseases where herbal medicine is most frequently used. The low prevalence of drug-induced liver injury (DILI) gives rise to the need for large-scale patient studies. The objective of this study is to report on the incidence of liver injury from herbal medicine in musculoskeletal disease patients as large-scale studies are scarce.

Of 32,675 inpatients taking herbal medicine at 7 locations of a Korean medicine hospital between 2005 and 2013, we screened for liver injury in 6,894 patients with liver function tests (LFTs) at admission and discharge. LFTs included t-bilirubin, AST, ALT, and ALP. We assessed for risk factors for liver injury at discharge.

Participants received the most frequently used complementary and alternative medicine treatment contents (herbal medicine, acupuncture, pharmacopuncture, bee venom pharmacopuncture, and Chuna manipulation) administered to musculoskeletal disease patients at this hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted for at least one day who took herbal medicine and at least 2 LFTs during admittance.

Exclusion Criteria:

* None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Musculoskeletal patients admitted to an integrated hospital that offers both complementary and alternative medicine (CAM) and conventional medicine treatment.
Sampling Method: Non-Probability Sample
Enrollment: 6894 (Actual)
Dates: Start 2005-12 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Alanine aminotransferase (ALT) | Change from baseline (admission) in liver function test up to discharge (average 4 wks)
  Participants were followed for the duration of hospital stay, an average of 4 weeks.
Aspartate aminotransferase (AST) | Change from baseline (admission) in liver function test up to discharge (average 4 wks)
  Participants were followed for the duration of hospital stay, an average of 4 weeks.
Alkaline phosphatase (ALP) | Change from baseline (admission) in liver function test up to discharge (average 4 wks)
  Participants were followed for the duration of hospital stay, an average of 4 weeks.
Total bilirubin (TB) | Change from baseline (admission) in liver function test up to discharge (average 4 wks)
  Participants were followed for the duration of hospital stay, an average of 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Jinho Lee, Masters, Principal Investigator — Jaseng Hospital of Korean Medicine
Locations (1):
- Jaseng Hospital of Korean Medicine, Seoul, Gangnam-Gu, South Korea